CLINICAL TRIAL: NCT07407829
Title: Step by Step Back - A Feasibility Study of a CBT-Based Physical Activity Intervention for Stress-Related Exhaustion
Brief Title: Step by Step Back - A Feasibility Study of a Physical Activity Intervention for Adults With Stress-related Exhaustion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: Itrim (Unknown); Avonova (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-04555-01
Record Dates: First submitted 2025-12-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Exhaustion Disorder; Stress-Related Disorders
Keywords: Stress-related exhaustion; Exhaustion disorder; Fatigue; Burnout; Physical activity intervention; Exercise therapy; Feasibility study; Cognitive behavioral therapy (CBT); Acceptance and Commitment Therapy (ACT); Psychological flexibility
MeSH Terms: conditions — Fatigue; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Single-group, open-label interventional mixed-methods feasibility study evaluating a clinician-guided physical activity program integrated into psychological treatment as usual for adults experiencing stress-related exhaustion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Clinician-guided physical activity program integrated into treatment as usual (Experimental): Participants receive a clinician-guided physical activity program integrated into regular psychological treatment as usual. The program is manualized and individually tailored to support gradual and sustainable engagement in physical activity. It is designed to be integrated into approximately 5 to 6 individual sessions delivered by a licensed psychologist or psychotherapist over a flexible time period depending on the participant's pace and circumstances.
  Interventions: Behavioral: CBT/ACT-based psychologist-delivered physical activity program

INTERVENTIONS:
Behavioral: CBT/ACT-based psychologist-delivered physical activity program — A structured psychologist-delivered physical activity program integrating Cognitive Behavioral Therapy (CBT) and Acceptance and Commitment Therapy (ACT) principles. It supports individuals with stress-related exhaustion in developing sustainable and value-based ways of being physically active. Core components include psychoeducation about fatigue and recovery, clarification of personal values, goal setting, and graded behavioral activation tailored to individual needs.
  The program consists of approximately 5-6 individual sessions, delivered by licensed psychologists over a flexible time period depending on the participant's pace and circumstances. Each session covers key themes such as understanding exhaustion and physical activity, identifying barriers and values, planning and adjusting activity, addressing unhelpful thoughts and emotions, and a flexible approach to physical activity (e.g. mode, frequency, duration, intensity). Between sessions, participants complete home exercises.

SUMMARY:
The goal of this clinical study is to learn whether a psychologist- or psychotherapist-guided physical activity program can be delivered and used as part of regular care for adults experiencing stress-related exhaustion. The program is designed to be integrated into regular psychological treatment as usual and supports participants in developing physical activity habits in a gradual, individualized, and sustainable way.

The main questions this study aims to answer are:

* Can participants complete the program and attend the planned sessions?
* Do participants and clinicians find the program acceptable, relevant, and useful?
* Is the program safe, and do any negative experiences occur during the program?
* What practical barriers and facilitators affect participation and delivery in routine care?
* What descriptive patterns of change are seen in physical activity, symptoms, and everyday functioning from before to after the program?

The program is based on cognitive behavioral therapy (CBT) and acceptance and commitment therapy (ACT). It includes strategies to help participants set meaningful goals, take step-by-step actions toward those goals, and respond more flexibly to uncomfortable thoughts, emotions, and body sensations that may arise in relation to physical activity.

About 12 to 20 participants will take part. The program is designed to be integrated into about 5 to 6 individual sessions delivered over a flexible time period, depending on each participant's pace and circumstances.

Participants will:

* Take part in the physical activity program as part of their regular psychological treatment
* Complete online questionnaires before and after the program
* Log their physical activity during the program
* Provide feedback after the program (and some participants will also take part in an interview)

The results will be used to assess whether the program is feasible and acceptable for participants and clinicians and to inform further refinement and future evaluation.

DETAILED DESCRIPTION:
Background and rationale Prolonged psychosocial stress can lead to substantial exhaustion, often accompanied by impaired cognitive function, sleep disturbance, and reduced everyday functioning. In Sweden, these difficulties have often been described within the diagnosis exhaustion disorder (ED), introduced in 2003 (International Classification of Diseases, 10th Revision, Swedish adaptation; ICD-10-SE F43.8A). ED is associated with high rates of sick leave and substantial societal costs. With the transition to the World Health Organization (WHO) International Classification of Diseases, 11th Revision (ICD-11), this national diagnosis will be phased out in 2028; however, the clinical problems it captures are expected to remain prevalent. There is therefore a need to continue developing and evaluating feasible and scalable rehabilitation approaches for individuals experiencing stress-related exhaustion.

Physical activity has well-documented preventive and rehabilitative effects on mental health problems such as depression, anxiety, and stress, but its role in rehabilitation for stress-related exhaustion has been less studied. In clinical practice, physical activity may be approached with caution in this group, and treatment recommendations have often emphasized rest and low-intensity activity. Many individuals struggle to reintroduce activity in a sustainable way: some avoid activity due to fear of symptom worsening, while others push themselves too hard. Over time, both patterns may contribute to persistent fatigue and reduced functioning.

A psychologically informed and individually tailored approach to graded physical activity may help participants develop a more sustainable activity pattern by supporting pacing and gradual progression, addressing avoidance and overexertion patterns, and strengthening engagement in meaningful life domains.

Intervention framework and development The intervention was developed within a broader research program on physical activity in stress-related exhaustion, including an experimental study on responses to acute exercise and a qualitative interview study on experiences and perceptions of physical activity during rehabilitation. Findings from these studies informed the content and delivery procedures of the present intervention.

The intervention is grounded in cognitive behavioral therapy (CBT) and acceptance and commitment therapy (ACT) principles and draws on established behavior change theories, including Social Cognitive Theory and dual-process models. Key processes targeted include self-efficacy, behavioral activation, and psychological flexibility. The intervention aims to support sustainable behavior change through values clarification, behavioral strategies, and gradual exposure to activity-related discomfort.

In line with guidance from the United Kingdom Medical Research Council (MRC) framework for developing and evaluating complex interventions, the present study is an early-stage evaluation focused on feasibility and acceptability. Findings will inform intervention refinement and planning of future evaluation.

Study design and setting This is a single-arm interventional feasibility study conducted in routine clinical care. All participants receive the intervention; there is no control or comparator arm. The program is delivered by licensed psychologists and psychotherapists and is designed to be integrated into regular psychological treatment as usual in clinical settings where stress-related exhaustion is commonly treated, including occupational health care and primary care. No masking is applied (open label), and allocation is not applicable.

A mixed-methods design is used to evaluate feasibility and explore participant and clinician experiences. Quantitative and qualitative data are collected in parallel and integrated during interpretation.

Participants and recruitment Adults meeting the protocol inclusion and exclusion criteria will be recruited consecutively via collaborating clinicians. The target sample size is approximately 12-20 participants, consistent with feasibility study guidance aimed at assessing acceptability, practicality, and safety and informing refinement of the intervention and study procedures.

Intervention description The intervention is a manualized CBT-based physical activity program integrated into psychological treatment as usual. It is individually tailored and structured to support participants in building sustainable physical activity habits through values-based work, behavioral strategies, and gradual progression.

The program acknowledges that individuals experiencing stress-related exhaustion may differ in functional profile and activity patterns. Some may avoid activity due to fear of symptom worsening or relapse, while others may struggle with overexertion. The intervention therefore emphasizes individualized pacing and progression and supports participants in responding flexibly to internal experiences such as fatigue-related sensations, thoughts, and emotions that may arise before, during, or after physical activity.

Key components include:

* Psychoeducation about fatigue and recovery processes and the role of physical activity from behavioral and learning-based perspectives
* Values clarification to support engagement in personally meaningful life domains
* Goal setting and action planning using graded task assignment and stepwise progression
* Graded exposure to physical activity, adapted to individual capacity and functional status
* Skills for responding flexibly to unhelpful thoughts and emotions related to physical activity, fatigue, performance, and relapse concerns
* Reflection on activity experiences, including affective responses, to support learning and motivation

The program is designed to be integrated into approximately 5-6 individual sessions delivered over a flexible time period depending on the participant's pace and circumstances. Brief home tasks are included between sessions.

Data collection procedures Quantitative and qualitative data are collected to evaluate feasibility and acceptability and to inform refinement of the intervention and study procedures.

Participants complete digital self-report questionnaires at baseline (approximately 1 week before program start) and post-intervention (approximately 1 week after program completion). During the intervention period, participants provide brief monitoring data related to physical activity engagement (date, duration, type of activity, rating of perceived exertion [RPE]) .

After completing the intervention, participants provide structured feedback about their experiences, and a subset participate in semi-structured interviews to explore perceived helpful and hindering aspects, barriers and facilitators, and suggestions for improvement. Psychologists and psychotherapists delivering the program also complete structured feasibility-related documentation to support evaluation of delivery and implementation in routine care.

To capture other potentially relevant care received during the intervention period, participants complete a brief post-intervention questionnaire on health care utilization adapted from the Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TIC-P). These data are collected to contextualize feasibility findings and descriptive outcome patterns rather than as a treatment outcome.

Feasibility focus and outcomes reporting The primary purpose of the study is to evaluate whether the intervention and study procedures are feasible and acceptable in primarily by adults with stress-related exhaustion, and also by clinicians in routine clinical settings. Feasibility is assessed using multiple pre-specified indicators, including intervention completion, attendance, adherence to intervention activities, fidelity of delivery, acceptability, and safety. These indicators are specified as separate outcome measures in the ClinicalTrials.gov record. Overall conclusions regarding feasibility will be based on combined interpretation of quantitative indicators and qualitative feedback.

In addition, descriptive pre-post patterns in participant-reported outcomes will be examined to support intervention refinement and planning of future evaluation (specified as separate outcome measures in the ClinicalTrials.gov record). The study is not designed or powered to provide confirmatory evidence of effectiveness.

Safety monitoring Safety is monitored throughout the intervention period. Any reported or observed adverse experiences (physical or psychological) are documented by the treating psychologist or psychotherapist. Participant feedback collected post-intervention is used to supplement safety documentation and capture experiences that may not have been reported during sessions.

Data analysis and mixed methods integration Quantitative data will be summarized using descriptive statistics. Exploratory analyses may be conducted to describe patterns of change and potential covariates using repeated-measures approaches, recognizing that the sample size is limited and that analyses are not confirmatory.

Qualitative interview data will be analyzed using thematic analysis, with inductive coding and theme development to capture participant experiences, perceived helpful and hindering aspects, and suggestions for refinement.

Quantitative and qualitative data will be analyzed separately and integrated at interpretation using joint displays and triangulation. Integration will be used to identify convergence, complementarity, and discrepancies across data sources to inform refinement of the intervention and support planning of future evaluation.

Progression considerations Decisions about further evaluation will primarily be informed by feasibility indicators and qualitative feedback on burden, fit, and perceived usefulness of the intervention. Findings will be used to refine the intervention and inform the design of a future larger-scale study.

ELIGIBILITY:
Inclusion Criteria

* Adult aged 20 to 64 years.
* Experiencing stress-related exhaustion, assessed in regular clinical care (for example, symptoms consistent with exhaustion disorder or a closely related stress-related condition).
* Symptoms are not in the acute phase (participant is able to engage in outpatient psychological treatment and gradual physical activity).
* Elevated fatigue/exhaustion at screening, indicated by scores on screening questionnaires (Karolinska Exhaustion Disorder Scale and Multidimensional Fatigue Inventory).
* Able to understand spoken and written Swedish.
* Has access to a smartphone, tablet, or computer with an internet connection to complete study questionnaires and activity logging.
* No medical condition that makes physical activity unsafe, based on clinical screening and participant self-report.

Exclusion Criteria

* Currently receiving psychological treatment outside the recruiting clinic that is expected to interfere with participation in the program or study assessments.
* Current or past diagnosis of a psychotic disorder.
* Current or past diagnosis of bipolar disorder.
* Severe mental health condition requiring another primary treatment approach at this time (for example, severe major depressive disorder, post-traumatic stress disorder, or an eating disorder).
* Ongoing substance use disorder.
* Medical condition or acute illness that makes physical activity inappropriate at this time (for example, recent blood clot, severe infection, or other serious condition).
* Severe musculoskeletal condition that substantially limits ability to perform physical activity.
* Started antidepressant medication within the past 4 weeks.

Additional notes (not eligibility criteria):

Participants may use psychotropic medication (for example, antidepressants, sleep medication, or anxiety medication) if the medication regimen is stable. Participants will be asked to report any medication changes during the study period. Mild to moderate comorbid anxiety or depression is allowed if stress-related exhaustion is the primary clinical problem.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Intervention completion (retention) | Up to 6 months
  Feasibility of the intervention will be primarily assessed by the proportion of participants who complete the intervention, defined as receiving a minimum dose of the program (attending at least 4 out of 6 intervention sessions delivered by a licensed psychologist or psychotherapist).

SECONDARY OUTCOMES:
Session attendance (intervention dose received) | Throughout the intervention period (from first to last session; approximately 5-6 sessions delivered over a flexible time period, typically within about 2-6 months).
  Attendance will be assessed as the number of intervention sessions attended during the program, recorded by the treating clinician (licensed psychologist or psychotherapist).
Participant adherence to intervention activities (home tasks and physical activity) | Throughout the intervention period (from first to last session; approximately 5-6 sessions delivered over a flexible time period, typically within about 2-6 months).
  Adherence will be assessed through clinician-recorded completion of assigned home exercises and through participant-reported physical activity engagement in the weekly activity log.
Intervention fidelity (delivery according to protocol) | Throughout the intervention period (from first to last session; approximately 5-6 sessions delivered over a flexible time period, typically within about 2-6 months).
  Fidelity will be assessed using clinicians' structured self-report documentation of delivered intervention components, recorded using a session documentation template and compared with the intended intervention protocol.
Safety (adverse events) | Throughout the intervention period (from first to last session; approximately 5-6 sessions delivered over a flexible time period, typically within about 2-6 months) and post-program questionnaires approximately 1 week after program cessation.
  Safety will be assessed by documentation of any reported or observed adverse events (physical or psychological) during the intervention period by the treating clinician (licensed psychologist or psychotherapist), and by self-report in post-program questionnaire. Reasons for discontinuation will be documented to identify any adverse-event-related attrition.
Participant acceptability and perceived fit (mixed methods) | Post-intervention (at intervention completion; after approximately 5-6 sessions delivered over a flexible time period, typically within about 2-6 months).
  Acceptability will be assessed using a brief post-intervention participant feedback questionnaire addressing perceived relevance, helpful and hindering aspects, missing components, perceived changes, and overall experience. A subset of participants will also complete a semi-structured interview based on the Change Interview protocol to provide more detailed qualitative feedback on acceptability, fit, barriers and facilitators, and suggestions for improvement.
Exhaustion symptoms (Karolinska Exhaustion Disorder Scale; KEDS) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in exhaustion symptoms measured with the Karolinska Exhaustion Disorder Scale (KEDS) total score (range 0-54; higher scores indicate greater exhaustion).
Fatigue (Multidimensional Fatigue Inventory; MFI-20) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in fatigue measured with the Multidimensional Fatigue Inventory (MFI-20) total score (range 20-100; higher scores indicate greater fatigue).
Burnout symptoms (Shirom-Melamed Burnout Measure; SMBM-12) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in burnout symptoms measured with the Shirom-Melamed Burnout Measure (SMBM-12) total score (mean score range 1-7; higher scores indicate greater burnout symptoms).
Anxiety symptoms (Hospital Anxiety and Depression Scale; HADS-A) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in anxiety symptoms measured with the Hospital Anxiety and Depression Scale, Anxiety subscale (HADS-A) score (range 0-21; higher scores indicate more anxiety symptoms).
Depressive symptoms (Hospital Anxiety and Depression Scale; HADS-D) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in depressive symptoms measured with the Hospital Anxiety and Depression Scale, Depression subscale (HADS-D) score (range 0-21; higher scores indicate more depressive symptoms).
Functional impairment (Work and Social Adjustment Scale; WSAS) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in functional impairment measured with the Work and Social Adjustment Scale (WSAS) total score (range 0-40; higher scores indicate greater functional impairment).
Psychological inflexibility related to fatigue (Psychological Inflexibility in Fatigue Scale; PIFS) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in psychological inflexibility related to fatigue measured with the Psychological Inflexibility in Fatigue Scale (PIFS) total score (12 items; range 0-84). Higher scores indicate greater fatigue-related avoidance and cognitive fusion (greater psychological inflexibility).
Exercise self-efficacy (Swedish Exercise Self-Efficacy Scale; S-ESES) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in exercise self-efficacy measured with the Swedish Exercise Self-Efficacy Scale (S-ESES) total score (10 items; range 10-40). Higher scores indicate greater confidence in ability to engage in physical activity/exercise.
Physical activity level (International Physical Activity Questionnaire; IPAQ) | Baseline and end of intervention (up to 6 months)
  Exploratory descriptive assessment of change in self-reported physical activity measured using the International Physical Activity Questionnaire (IPAQ) (reported using standard scoring; higher values indicate higher physical activity).
Weekly physical activity behavior (activity log) | From 1 week before the first intervention session through 1 week after the final intervention session.
  Exploratory descriptive assessment of physical activity behavior during the intervention period using weekly participant-reported activity logs capturing type of activity and duration. The primary descriptive variable will be total minutes of physical activity per week (higher values indicate more physical activity).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Blom, Professor, Principal Investigator — Department of Physical Activity and Health, The Swedish School of Sport and Health Sciences, Stockholm, Sweden.
Locations (1):
- Avonova Occupational Health, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The data analyzed or produced in this study will not be openly accessible due to Swedish legislation (the Swedish Ethical Review Act: 2003:460) but the authors can provide access upon reasonable request. For such inquiries, please contact Victoria Blom, victoria.blom@gih.se.

REFERENCES:
- [Background] Braun V, Clarke, V. Thematic Analysis: A Practical Guide. Sage Publications; 2021.
- [Background] Elliott R, Slatick E, Urman M. Qualitative change process research on psychotherapy: alternative strategies. Psychol Test Assess Model. (2001) 43:69.
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Timman R, Bouwmans C, Busschbach JJ, Hakkaart-van Roijen L. Development of the Treatment Inventory of Costs in Psychiatric Patients: TIC-P Mini and Midi. Value Health. 2015 Dec;18(8):994-9. doi: 10.1016/j.jval.2015.07.006. Epub 2015 Sep 16. PMID 26686783
- [Background] Russel JA. A circumplex model of affect. J. Pers. Soc. Psychol. 1980; 39(6):1161-1178.
- [Background] Beauchaine TP, Thayer JF. Heart rate variability as a transdiagnostic biomarker of psychopathology. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):338-350. doi: 10.1016/j.ijpsycho.2015.08.004. Epub 2015 Aug 11. PMID 26272488
- [Background] Tiwari R, Kumar R, Malik S, Raj T, Kumar P. Analysis of Heart Rate Variability and Implication of Different Factors on Heart Rate Variability. Curr Cardiol Rev. 2021;17(5):e160721189770. doi: 10.2174/1573403X16999201231203854. PMID 33390146
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Ahlstrom I, Hellstrom K, Emtner M, Anens E. Reliability of the Swedish version of the Exercise Self-Efficacy Scale (S-ESES): a test-retest study in adults with neurological disease. Physiother Theory Pract. 2015 Mar;31(3):194-9. doi: 10.3109/09593985.2014.982776. Epub 2014 Nov 24. PMID 25418018
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Saltin B, Grimby G. Physiological analysis of middle-aged and old former athletes. Comparison with still active athletes of the same ages. Circulation. 1968 Dec;38(6):1104-15. doi: 10.1161/01.cir.38.6.1104. No abstract available. PMID 5721960
- [Background] Lundqvist J, Lindberg MS, Brattmyr M, Havnen A, Hjemdal O, Solem S. The Work and Social Adjustment Scale (WSAS): An investigation of reliability, validity, and associations with clinical characteristics in psychiatric outpatients. PLoS One. 2024 Oct 10;19(10):e0311420. doi: 10.1371/journal.pone.0311420. eCollection 2024. PMID 39388411
- [Background] Jonsjö MA, Wicksell RK, Holmström L, , Andreasson A, Olsson GL. Acceptance & Commitment Therapy for ME/CFS (Chronic Fatigue Syndrome) - A feasibility study. J. Context. Behav. Sci. 2019 Apr;12:89-97.
- [Background] Wicksell RK, Renofalt J, Olsson GL, Bond FW, Melin L. Avoidance and cognitive fusion--central components in pain related disability? Development and preliminary validation of the Psychological Inflexibility in Pain Scale (PIPS). Eur J Pain. 2008 May;12(4):491-500. doi: 10.1016/j.ejpain.2007.08.003. Epub 2007 Sep 20. PMID 17884643
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Beser A, Sorjonen K, Wahlberg K, Peterson U, Nygren A, Asberg M. Construction and evaluation of a self rating scale for stress-induced exhaustion disorder, the Karolinska Exhaustion Disorder Scale. Scand J Psychol. 2014 Feb;55(1):72-82. doi: 10.1111/sjop.12088. Epub 2013 Nov 15. PMID 24236500
- [Background] Åsberg M, editor. Utmattningssyndrom. 1st ed. Stockholm: Gothia Kompetens; 2024.
- [Background] Almén N, Jansson B. The reliability and factorial validity of different versions of the Shirom-Melamed Burnout Measure/Questionnaire and normative data for a general Swedish sample. Int J Stress Manag. 2021;28(4):314-325
- [Background] Hagelin CL, Wengstrom Y, Runesdotter S, Furst CJ. The psychometric properties of the Swedish Multidimensional Fatigue Inventory MFI-20 in four different populations. Acta Oncol. 2007;46(1):97-104. doi: 10.1080/02841860601009430. PMID 17438711
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. Int J Nurs Stud. 2024 Jun;154:104705. doi: 10.1016/j.ijnurstu.2024.104705. Epub 2024 Feb 24. PMID 38564982
- [Background] Hofmann SG, Asmundson GJ, Beck AT. The science of cognitive therapy. Behav Ther. 2013 Jun;44(2):199-212. doi: 10.1016/j.beth.2009.01.007. Epub 2011 May 25. PMID 23611069
- [Background] Choi J, Lee M, Lee JK, Kang D, Choi JY. Correlates associated with participation in physical activity among adults: a systematic review of reviews and update. BMC Public Health. 2017 Apr 24;17(1):356. doi: 10.1186/s12889-017-4255-2. PMID 28438146
- [Background] Hayes SC, Strosahl KD, Wilson KG. ACT Acceptance and Commitment Therapy i teori och tillämpning: Vägen till psykologisk flexibilitet. 2. Uppl. Ruthman M. Stockholm: Natur & Kultur; 2014.
- [Background] Brand R, Ekkekakis P. Affective-reflective theory of physical inactivity and exercise. Ger J Exerc Sport Res. 2018:48(1);48-58.
- [Background] Biddle S, Mutrie N, Gorely T, Faulkner G. Psychology of Physical Activity: Determinants, Well-Being and Interventions. 4th ed. New York and London: Routledge; 2021.
- [Background] The Swedish Social Insurance Agency (2020). Sickness absence in psychiatric disorders (Sjukfrånvaro i psykiatriska diagnoser)
- [Background] Åsberg M, Herlofsen J, Glise K. (2003). Utmattningssyndrom. Stressrelaterad psykisk ohälsa. Socialstyrelsen.
- [Background] Gerber M, Jonsdottir IH, Arvidson E, Lindwall M, Lindegard A. Promoting graded exercise as a part of multimodal treatment in patients diagnosed with stress-related exhaustion. J Clin Nurs. 2015 Jul;24(13-14):1904-15. doi: 10.1111/jocn.12820. Epub 2015 May 4. PMID 25939917
- [Background] Eskilsson T, Slunga Jarvholm L, Malmberg Gavelin H, Stigsdotter Neely A, Boraxbekk CJ. Aerobic training for improved memory in patients with stress-related exhaustion: a randomized controlled trial. BMC Psychiatry. 2017 Sep 2;17(1):322. doi: 10.1186/s12888-017-1457-1. PMID 28865430
- [Background] Lindegard A, Jonsdottir IH, Borjesson M, Lindwall M, Gerber M. Changes in mental health in compliers and non-compliers with physical activity recommendations in patients with stress-related exhaustion. BMC Psychiatry. 2015 Nov 4;15:272. doi: 10.1186/s12888-015-0642-3. PMID 26530329
- [Background] Noetel M, Sanders T, Gallardo-Gomez D, Taylor P, Del Pozo Cruz B, van den Hoek D, Smith JJ, Mahoney J, Spathis J, Moresi M, Pagano R, Pagano L, Vasconcellos R, Arnott H, Varley B, Parker P, Biddle S, Lonsdale C. Effect of exercise for depression: systematic review and network meta-analysis of randomised controlled trials. BMJ. 2024 Feb 14;384:e075847. doi: 10.1136/bmj-2023-075847. PMID 38355154
- [Background] Oslo Chronic Fatigue Consortium; Alme TN, Andreasson A, Asprusten TT, Bakken AK, Beadsworth MB, Boye B, Brodal PA, Brodwall EM, Brurberg KG, Bugge I, Chalder T, Due R, Eriksen HR, Fink PK, Flottorp SA, Fors EA, Jensen BF, Fundingsrud HP, Garner P, Havdal LB, Helgeland H, Jacobsen HB, Johnson GE, Jonsjo M, Knoop H, Landmark L, Launes G, Lekander M, Linnros H, Lindsater E, Liira H, Linnestad L, Loge JH, Lyby PS, Malik S, Malt UF, Moe T, Norlin AK, Pedersen M, Pignatiello SE, Rask CU, Reme SE, Roksund G, Sainio M, Sharpe M, Thorkildsen RF, van Roy B, Vandvik PO, Vogt H, Wyller HB, Wyller VBB. Chronic fatigue syndromes: real illnesses that people can recover from. Scand J Prim Health Care. 2023 Dec;41(4):372-376. doi: 10.1080/02813432.2023.2235609. Epub 2023 Nov 29. PMID 37740918
- [Background] Lindsater E, Svardman F, Rosquist P, Wallert J, Ivanova E, Lekander M, Soderholm A, Ruck C. Characterization of exhaustion disorder and identification of outcomes that matter to patients: Qualitative content analysis of a Swedish national online survey. Stress Health. 2023 Oct;39(4):813-827. doi: 10.1002/smi.3224. Epub 2023 Jan 27. PMID 36645034
- [Background] Kling J, Persson Asplund R, Ekblom O, Blom V. Psychological responses to acute exercise in patients with stress-induced exhaustion disorder: a cross-over randomized trial. BMC Psychiatry. 2025 Jan 24;25(1):72. doi: 10.1186/s12888-025-06484-1. PMID 39856671
- [Background] Lindsater E, Svardman F, Wallert J, Ivanova E, Soderholm A, Fondberg R, Nilsonne G, Cervenka S, Lekander M, Ruck C. Exhaustion disorder: scoping review of research on a recently introduced stress-related diagnosis. BJPsych Open. 2022 Aug 24;8(5):e159. doi: 10.1192/bjo.2022.559. PMID 36458830
- [Background] Loy BD, O'Connor PJ, Dishman RK. The effect of a single bout of exercise on energy and fatigue states: a systematic review and meta-analysis. Fatigue. 2013;1(4):223-242.
- [Background] Mikkelsen K, Stojanovska L, Polenakovic M, Bosevski M, Apostolopoulos V. Exercise and mental health. Maturitas. 2017 Dec;106:48-56. doi: 10.1016/j.maturitas.2017.09.003. Epub 2017 Sep 7. PMID 29150166
- [Background] Singh B, Olds T, Curtis R, Dumuid D, Virgara R, Watson A, Szeto K, O'Connor E, Ferguson T, Eglitis E, Miatke A, Simpson CE, Maher C. Effectiveness of physical activity interventions for improving depression, anxiety and distress: an overview of systematic reviews. Br J Sports Med. 2023 Sep;57(18):1203-1209. doi: 10.1136/bjsports-2022-106195. Epub 2023 Feb 16. PMID 36796860